CLINICAL TRIAL: NCT06362447
Title: Phase 2 Study Evaluating the Efficacy of Injectable Gentamicin in Hereditary Ichthyosis
Brief Title: Efficacy of Injectable Gentamicin in Hereditary Ichthyosis
Acronym: GENTIC
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RC31/22/0320
Record Dates: First submitted 2024-04-02; First posted 2024-04-12 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2024-08

CONDITIONS: Ichthyosis
Keywords: Congenital ichthyoses; injectable gentamicin
MeSH Terms: conditions — Ichthyosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Gentamicin (Experimental): Gentamicin injection
  Interventions: Drug: Gentamicin Injectable Solution

INTERVENTIONS:
Drug: Gentamicin Injectable Solution — Gentamicin (10 mg/kg) will be administrated once weekly for 3 months

SUMMARY:
This study will evaluate the efficacy and safety of intravenous gentamicin in congenital ichthyosis due to a non-sens mutation. The primary objective is the severity of scales and erythema at the third month, compared to baseline. Secondary objectives will include: the importance of itching, trans epidermal water loss, cutaneous expression of the targeted protein, the security of the drug and patients' satisfaction.

DETAILED DESCRIPTION:
Congenital ichthyoses represent a group of diseases characterized by disabling cutaneous anomalies (scales and inconstant erythema) often associated with extra cutaneous anomalies that may be severe. The treatment is non curative and symptomatic, including local treatments (ie. emollients). Oral retinoids may be helpful in moderate to severe forms. There is a huge need for novel therapies, ideally targeting the molecular defect. Gentamicin may be a novel therapeutic option for congenital ichthyosis.

Apart its antimicrobial effect, gentamicin can achieve stop codon readthrough and produce full-length protein.

In this study, gentamicin (10 mg/kg) will be administrated once weekly for 3 months. The study will include monthly visits, a follow-up visit 3 months after the stopping the drug and an end-of-study visit 3 months after the follow-up visit. Kidney and hearing functions will be assessed regularly.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients affiliated to a social insurance protection regimen.
2. Hereditary ichthyosis caused by a homozygous non-sense mutation of a gene responsible for hereditary ichthyosis (TGM1, PNPLA1, ALOX12B, NIPAL4, ALOXE3, SDR9C7, ABCA12, CERS3, SPINK5 and CDSN)
3. Moderate to severe forms of ichthyosis defined as Validating an Ichthyosis Severity Index score at 2-3 on at least 2 out of 4 areas evaluated (back, upper limbs, lower limbs, back of the foot)
4. Free, informed consent, written and signed by the participant and the investigator (at the latest on the day of inclusion and before any examination required by the research).

Exclusion Criteria:

1. Cutaneous signs suggesting a surinfection
2. Hypersensibility of active substance or one of the gentamicin excipients
3. Administration of an aminoside in the previous 3 months
4. Treatment with nephrotoxic or ototoxic medication in the previous 6 weeks
5. Pregnant or breastfeeding women, or women planning to become pregnant or breastfeed during the study. Women of childbearing age, potentially sexually active, and unwilling to use acceptable contraception measures in accordance with Clinical Trials Facilitation and Coordination Group recommendations
6. Subjects >75 years (physiological impairment of kidney function)
7. Left ventricular insufficiency
8. Hypoalbuminemia
9. Myasthenia
10. History of necrosis at the injection site during previous treatment with aminosid
11. Grade B or C cirrhosis according to Child-Pugh classification
12. Nephropathy or other situation at risk of renal dysfunction
13. Renal insufficiency with glomerular filtration rate < 60mL/min
14. Surdity which is not caused by plug scales in the external ear canals or other situation at risk of surdity including the presence of the A1555G mutation in the 12S ribonucleic acid (mitochondrial deoxyribonucleic acid) gene
15. Patient who modify his keratolytic or emollient treatment in the last two weeks previous the inclusion visit
16. Patient who modify his retinoid topic treatment in the month previous the inclusion visit
17. Patient who modify his systemic retinoid treatment in the 3 months previous the inclusion visit
18. Patient under guardianship, curatorship or deprived of their liberty
19. Patient with pre-existing neuromuscular disease
20. Patient participating in another clinical study with investigational treatment

Exclusion criteria at the end of the "run-in" period:

Variation greater than 15% in the Validating an Ichthyosis Severity Index score between two baseline measurements.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Gentamicin efficacity | 3 months
  Proportion of patients with a reduction in Visual Index of Ichthyosis Severity score of at least 15%

SECONDARY OUTCOMES:
Gentamicin efficacity | Month 1, Month 2, Month 4, Month 5, Month 6 and Month 9
  Proportion of patients with a reduction in Visual Index of Ichthyosis Severity score
Gentamicin efficacity on quality of life | Month 3, Month 6 and Month 9
  Assessment of quality of life by IQoL-32 score (specific to ichthyosis)

CONTACTS AND LOCATIONS:
Overall Officials: SEVERINO-FREIRE Maella, MD, Principal Investigator — University Hospital, Toulouse
Locations (2):
- France (2):
  - Hôpital Saint-Louis APHP, Paris, France
  - CHU de Toulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: No